CLINICAL TRIAL: NCT03635736
Title: Study on Additive Use of Non-invasive Acustocerebrography in Patients Suspect to Severe Brain Injury
Brief Title: Acustocerebrography (ACG) in Severe Brain Injury
Acronym: ACG-BrainICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dr. Martin Sauer, MD, PD. Dr. med. habil.; Deputy on Intensive Care Medicine, University of Rostock
Other Study IDs: A 2018-0062
Record Dates: First submitted 2018-07-25; First posted 2018-08-17 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Brain Injuries, Acute
Keywords: brain damage; sonography
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe brain injury: ICU-patients suspect to severe brain injury, measurement with multiple-spectral-sonography as acustocerebrography (ACG
  Interventions: Other: multiple-spectral-sonography as acustocerebrography (ACG)

INTERVENTIONS:
Other: multiple-spectral-sonography as acustocerebrography (ACG) — After inclusion three times at day measurements with ACG for each 45 minutes; a (non-invasive) sonography. The measurements will be stopped after final evaluation of the neurological status using common methods like magnetic resonance tomography, transcranial doppler sonography, electroencephalography and other methods.

SUMMARY:
The study will enable the clinical applicability of the multiple-spectral-sonography for detection of severe brain injury in ICU patients. For this, the ACG diagnostic system (Sonovum AG, Leipzig, Germany) should be used as additional diagnostic tool in prospective single-center study.

DETAILED DESCRIPTION:
A multiple-step procedure, including repetition of the clinical examinations after a waiting period and use of additional technical diagnostic tools e.g. magnetic resonance tomography and Transcranial Doppler sonography (TCD) are needed for determining of severe brain injury and irreversible brain function failure.

This study will enable the clinical applicability of the multiple-spectral-sonography for detection of severe brain injury in ICU patients. For this, the ACG diagnostic system (Sonovum AG, Leipzig, Germany) should be used as additional diagnostic tool in prospective single-center study.

The ACG-method is a bedside non-invasive sonography that has been shown to be useful in previous studies analyzing circulatory changes in rat cerebral blood vessels, for example, to distinguish between brain-ischemia and -hemorrhage. Additionally, in the case of brain death, the spontaneous electrical activity, which can be measured by means of ACG as global elasticity, was not longer detectable.

In the study should include 30 adult ICU-patients in patients suspect to severe brain injury. The inclusion of patients will be started if written informed consent was obtained from participants or their representatives. After the inclusion, the ACG is measured three times a day. In addition, the routinely practice (treatment and diagnostic) for patients with severe brain injury (neurological clinical examinations, use of additional technical diagnostic tools e.g. magnetic resonance tomography and Transcranial Doppler sonography (TCD); Standard Medical Care) should be made and documented. From all patients basic demographic data, pre-morbidity, vital parameters, blood parameters, Illness severity scores (APACHE-II, SOFA, GCS), drug levels, microbiological results and cranial MRI/CT results will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* suspected severe brain injury

Exclusion Criteria:

* open skull brain trauma
* skull fractures in the temporal area
* decompression-craniotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - ICU-patients over 17 years old with suspected severe brain injury
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
acustocerebrography (ACG) | after inclusion: time-point 0 hours
  changes in the ACG during the course of disease (especially the dimensionality of the time to flight of the ultrasound signal)

SECONDARY OUTCOMES:
SOFA | every day, at least after 28 days
  Evaluation of the SOFA-Score
acustocerebrography (ACG) | Every day to 3 time-points. The measurements will be stopped after final evaluation of the neurological status, at least after 28 days
  changes in the ACG during the course of disease (especially the dimensionality of the time to flight of the ultrasound signal)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sauer, MD, Principal Investigator — University Hospital of Rostock, Germany
Locations (1):
- Intensive Care Units PIT 1+2, University hospital Rostock, Rostock, Germany